CLINICAL TRIAL: NCT02778919
Title: Late Phase II Clinical Study of KLH-2109 in Patients With Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KLH1204
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — linzagolix; Leuprolide

ARMS (6):
- KLH-2109, lowest dose (Experimental)
  Interventions: Drug: KLH-2109; Drug: Placebo
- KLH-2109, low dose (Experimental)
  Interventions: Drug: KLH-2109; Drug: Placebo
- KLH-2109, medium dose (Experimental)
  Interventions: Drug: KLH-2109; Drug: Placebo
- KLH-2109, high dose (Experimental)
  Interventions: Drug: KLH-2109
- Placebo (Placebo Comparator): First 12 week period; Placebo, Second 12 week period; randomize to one of the KLH-2109 dose levels
  Interventions: Drug: Placebo
- Leuprorelin acetate (Other): Active reference
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: KLH-2109
  Arms: KLH-2109, high dose; KLH-2109, low dose; KLH-2109, lowest dose; KLH-2109, medium dose
Drug: Placebo
  Arms: KLH-2109, low dose; KLH-2109, lowest dose; KLH-2109, medium dose; Placebo
Drug: Leuprorelin acetate
  Arms: Leuprorelin acetate

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and dose-response relationship of KLH-2109 compared to placebo in Japanese patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with endometriosis

Exclusion Criteria:

* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Change of average Numerical Rating Scale (NRS) score of pelvic pain | 12 weeks

SECONDARY OUTCOMES:
Incidences of adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Japan